CLINICAL TRIAL: NCT01779570
Title: Anti-inflammatory Effects of Macrolide Treatment in Influenza Lower Respiratory Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Nelson Lee, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGC CUHK468112
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Influenza; Lower Respiratory Tract Infection
Keywords: Influenza; Macrolide; Anti-inflammatory
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macrolide treatment (Experimental): Azithromycin 500 mg daily for 5 days
  Interventions: Drug: Macrolide treatment
- No macrolide treatment (No Intervention): No azithromycin

INTERVENTIONS:
Drug: Macrolide treatment
  Arms: Macrolide treatment

SUMMARY:
Influenza lower respiratory tract infection (LRTI) is a major cause of morbidity and mortality worldwide. While viral replication can be suppressed by antiviral treatment, excessive inflammatory responses, which are increasingly recognized to contribute to severe influenza complications, remain unopposed. Macrolides have been used widely to treat community-acquired pneumonia, and shown to exert anti-inflammatory effects in other respiratory diseases, providing clinical benefits. In this randomized, open-label, multicenter study, we aim to investigate the anti-inflammatory effects of macrolide treatment in influenza LRTI. Its impacts on the cytokine response, viral clearance, symptoms and disease resolution will be studied. Such results may lead to the development of new therapeutic approaches against severe influenza infection, and provide better insights into disease pathogenesis.

DETAILED DESCRIPTION:
Objectives: (1) We aim to investigate the anti-inflammatory effects of macrolide treatment in patients with influenza LRTI and the impact on viral clearance. (2) To investigate the impact of macrolide treatment on influenza symptom and disease resolution.

Design: A randomized, open-label, multicenter study.

Settings: Acute medical facilities in 3 general public hospitals in Hong Kong.

Subjects, Sampling and Intervention: Adult (>/=18 years) patients hospitalized for virologically confirmed influenza LRTI who fulfill the inclusion/exclusion criteria will be randomized to receive (1) azithromycin 500 mg p.o. for 5 days (in addition to antiviral, as part of usual care), or (2) no azithromycin (ie, antiviral alone, part of usual care) after informed consent. Serial blood samples will be collected for cytokine/inflammatory response assays. Serial nasopharyngeal swabs will be collected to assess for viral clearance. Symptoms, clinical progress, radiography and adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. established influenza A or B infection by virologic tests
2. age >/=18 years
3. present within 4 days from illness onset
4. clinical evidence of LRTI and require hospital care
5. require antiviral (oseltamivir) treatment
6. able to provide written, informed consent.

Exclusion Criteria:

1. patients on immunosuppressants
2. pregnant or lactating woman
3. known hepatic failure, end-stage renal failure, cardiac arrhythmia (e.g. prolonged corrected QT interval >450 msec)
4. known contraindications to azithromycin (e.g. allergic reaction)
5. lack of consent for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
cytokine and inflammatory responses | within 10 days post-intervention
  Serial measurements of selected cytokines/chemokines (e.g. interleukin-6, CXCL8) and proinflammatory molecules (e.g. DAMPs)

SECONDARY OUTCOMES:
viral clearance | within 10 days post-intervention
  Viral RNA and culture negativity in serially collected respiratory tract specimens

OTHER OUTCOMES:
time to recovery | within 10 days post-intervention
  e.g. time to symptom resolution, time to hospital discharge, etc

CONTACTS AND LOCATIONS:
Overall Officials: Nelson LS Lee, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong

REFERENCES:
- [Background] Chan PK, Chan MC, Cheung JL, Lee N, Leung TF, Yeung AC, Wong MC, Ngai KL, Nelson EA, Hui DS. Influenza B lineage circulation and hospitalization rates in a subtropical city, Hong Kong, 2000-2010. Clin Infect Dis. 2013 Mar;56(5):677-84. doi: 10.1093/cid/cis885. Epub 2012 Oct 16. PMID 23074315
- [Background] Chan PK, Lee N, Zaman M, Adisasmito W, Coker R, Hanshaoworakul W, Gasimov V, Oner AF, Dogan N, Tsang O, Phommasack B, Touch S, Bamgboye E, Swenson A, Toovey S, Dreyer NA. Determinants of antiviral effectiveness in influenza virus A subtype H5N1. J Infect Dis. 2012 Nov;206(9):1359-66. doi: 10.1093/infdis/jis509. Epub 2012 Aug 20. PMID 22927451
- [Background] Lee N, Ison MG. Diagnosis, management and outcomes of adults hospitalized with influenza. Antivir Ther. 2012;17(1 Pt B):143-57. doi: 10.3851/IMP2059. Epub 2012 Feb 3. PMID 22311561
- [Background] Lee N, Wong CK, Chan PK, Chan MC, Wong RY, Lun SW, Ngai KL, Lui GC, Wong BC, Lee SK, Choi KW, Hui DS. Cytokine response patterns in severe pandemic 2009 H1N1 and seasonal influenza among hospitalized adults. PLoS One. 2011;6(10):e26050. doi: 10.1371/journal.pone.0026050. Epub 2011 Oct 13. PMID 22022504
- [Background] Lee N, Chan PK, Lui GC, Wong BC, Sin WW, Choi KW, Wong RY, Lee EL, Yeung AC, Ngai KL, Chan MC, Lai RW, Yu AW, Hui DS. Complications and outcomes of pandemic 2009 Influenza A (H1N1) virus infection in hospitalized adults: how do they differ from those in seasonal influenza? J Infect Dis. 2011 Jun 15;203(12):1739-47. doi: 10.1093/infdis/jir187. PMID 21606532
- [Background] Lee N, Chan PK, Wong CK, Wong KT, Choi KW, Joynt GM, Lam P, Chan MC, Wong BC, Lui GC, Sin WW, Wong RY, Lam WY, Yeung AC, Leung TF, So HY, Yu AW, Sung JJ, Hui DS. Viral clearance and inflammatory response patterns in adults hospitalized for pandemic 2009 influenza A(H1N1) virus pneumonia. Antivir Ther. 2011;16(2):237-47. doi: 10.3851/IMP1722. PMID 21447873
- [Background] Lee N, Choi KW, Chan PK, Hui DS, Lui GC, Wong BC, Wong RY, Sin WY, Hui WM, Ngai KL, Cockram CS, Lai RW, Sung JJ. Outcomes of adults hospitalised with severe influenza. Thorax. 2010 Jun;65(6):510-5. doi: 10.1136/thx.2009.130799. PMID 20522848
- [Background] Hui DS, Lee N, Chan PK. Clinical management of pandemic 2009 influenza A(H1N1) infection. Chest. 2010 Apr;137(4):916-25. doi: 10.1378/chest.09-2344. Epub 2009 Dec 18. PMID 20022969
- [Background] Lee N, Chan PK, Hui DS, Rainer TH, Wong E, Choi KW, Lui GC, Wong BC, Wong RY, Lam WY, Chu IM, Lai RW, Cockram CS, Sung JJ. Viral loads and duration of viral shedding in adult patients hospitalized with influenza. J Infect Dis. 2009 Aug 15;200(4):492-500. doi: 10.1086/600383. PMID 19591575
- [Background] Lee N, Wong CK, Chan PK, Lun SW, Lui G, Wong B, Hui DS, Lam CW, Cockram CS, Choi KW, Yeung AC, Tang JW, Sung JJ. Hypercytokinemia and hyperactivation of phospho-p38 mitogen-activated protein kinase in severe human influenza A virus infection. Clin Infect Dis. 2007 Sep 15;45(6):723-31. doi: 10.1086/520981. Epub 2007 Aug 8. PMID 17712756
- [Background] Lee N, Chan PK, Choi KW, Lui G, Wong B, Cockram CS, Hui DS, Lai R, Tang JW, Sung JJ. Factors associated with early hospital discharge of adult influenza patients. Antivir Ther. 2007;12(4):501-8. PMID 17668558
- [Derived] Lee N, Wong CK, Chan MCW, Yeung ESL, Tam WWS, Tsang OTY, Choi KW, Chan PKS, Kwok A, Lui GCY, Leung WS, Yung IMH, Wong RYK, Cheung CSK, Hui DSC. Anti-inflammatory effects of adjunctive macrolide treatment in adults hospitalized with influenza: A randomized controlled trial. Antiviral Res. 2017 Aug;144:48-56. doi: 10.1016/j.antiviral.2017.05.008. Epub 2017 May 20. PMID 28535933
- See also: Division of Infectious Diseases, Department of Medicine and Therapeutics, The Chinese University of Hong Kong — http://www.mect.cuhk.edu.hk/specialties/infectiousdiseases.html